CLINICAL TRIAL: NCT06630481
Title: Long-term Survival Outcomes According to the Pathologic Response After Neoadjuvant Treatment in PDAC and the Fate of the Patients with Good CAP Grade
Acronym: CAP with NAT
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Professor, Seoul National University Hospital
Other Study IDs: 2407-036-1558
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer; Neoadjuvant Therapy; Pathological Complete Response
Keywords: CAP grade; tumor response grading system
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- CAP grade 0: No viable cancer cells in pancreatic resection specimen with neoadjuvant therapy.
  Interventions: Drug: neoadjuvant therapy
- CAP grade 1: Single cells or rare small groups of cancer cells in pancreatic resection specimen with neoadjuvant therapy.
  Interventions: Drug: neoadjuvant therapy
- CAP grade 2: Residual cancer with evident tumor regression in pancreatic resection specimen with neoadjuvant therapy.
  Interventions: Drug: neoadjuvant therapy
- CAP grade 3: Extensive residual cancer with no evident tumor regression in pancreatic resection specimen with neoadjuvant therapy.
  Interventions: Drug: neoadjuvant therapy
- pathological complete response: No viable cancer cells in pancreatic resection specimen with neoadjuvant therapy.
  Interventions: Drug: neoadjuvant therapy

INTERVENTIONS:
Drug: neoadjuvant therapy — Neoadjuvant chemotherapy, neoadjuvant radiotherapy, or both.

SUMMARY:
1. Neoadjuvant treatment (NAT) is increasingly used in managing pancreatic ductal adenocarcinoma (PDAC), necessitating dependable methods to evaluate tumor response.
2. Among various pathological tumor regression grading systems, the College of American Pathologists (CAP) system is commonly used to predict chemo-responsiveness and survival.
3. This study aimed to analyze long-term survival outcomes based on pathologic response using the CAP grade after NAT in PDAC and to identify clinicopathologic factors that influence a favorable pathologic response.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged >18 years) who underwent pancreatic resection after NAT at a single center between January 2009 and December 2023.
* Patients were initiated on NAT after confirming PDAC diagnosis based on pathological examination.

Exclusion Criteria:

* Patients without a reported CAP grade
* Patients who underwent palliative surgery
* Patients who received NAT outside the specified protocol due to incomplete information.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients (aged >18 years) who underwent pancreatic resection after NAT at Seoul National University Hospital between January 2009 and December 2023 were included. Patients were initiated on NAT after confirming PDAC diagnosis based on pathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
5-year overall survival | assessed up to 60months
  from diagnosis to any cause of death
5-year disease-free survival | assessed up to 60months
  defined as the duration between the date of surgery and the occurrence of the first instance of recurrence, death, or the last follow-up date.